CLINICAL TRIAL: NCT04499495
Title: A Retrospective Study to Assess 5-Aminosalicylic Acid Prescription Patterns and Treatment Outcomes in Patients With Ulcerative Colitis in Korea
Brief Title: Assessment of 5-Aminosalicylic Acid Prescription Patterns and Treatment Outcomes in Patients With Ulcerative Colitis in Korea
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000388
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-05

CONDITIONS: Ulcerative Colitis
Keywords: Mesalamine; Retrospective; 5-aminosalicylic acid; Prescription pattern
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: PENTASA (mesalamine/ 5-Aminosalicylic acid (5-ASA) — The 5-ASAs of interest in the study are mesalazine (5-ASA); sulfasalazine (5-ASA+sulfapyridine); and balsalazide (5-ASA) and will be grouped together as 5-ASA. For sulfasalazine and balsalazide, the equivalent dose to 5-ASA will be calculated as: balsalazide 6.75g is equivalent to 2.4g of mesalamine; and Sulfasalazine 4g is equivalent to 1.6g of mesalamine.
  The dose will be stratified by oral monotherapy, rectal monotherapy, oral and rectal combination therapy.

SUMMARY:
The prevalence of ulcerative colitis (UC), which is one of the inflammatory bowel diseases, is known to be increasing and the majority of patients (≥ 85%) have experienced mild or moderate severity.

5-Aminosalicylic acid (5-ASA), immunomodulator, or biologics, etc are prescribed to treat UC, however 5-ASA is generally considered the first-line therapy. The recent UC treatment guideline in Korea and the United States/ European Union (US/EU) have recommended higher daily dose for patients with mild or moderate severity than the previous guidelines since 2017. Accordingly, it is assumed that the average daily treatment dose of 5-ASA would increase in patients who were initially diagnosed with UC in real-world clinical practice in Korea. However, there are not many studies evaluating the treatment patterns and health outcomes of 5-ASA based on the recent treatment guideline in South Korea.

This study, hence, aims to investigate the impact of changes in daily dose of 5-ASA on the treatment patterns and health outcomes such as recurrence rate, hospitalization rate, and surgery rate in real world practice using Health Insurance Review and Assessment (HIRA) claims database.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed with UC during the index period.
* Patients who had at least two claims of 5-ASA (sulfasalazine, balsalazide, mesalamine) during the index period.
* Patients who underwent at least one endoscopy within a 3-month period prior to the index date (i.e. the first date of diagnosis with UC).

  * Defined as a claim with relevant endoscopy procedure code.
  * Include the upper gastrointestinal endoscopy, colonoscopy, sigmoidoscopy, which are identified using the procedure code.
* Patients who were treated with 5-ASA continuously for at least 1-month after the index date.

  * Defined as those who were treated with 5-ASA for more than 30 days within 6-month after the index date (i.e. the first date of diagnosis with UC).

Exclusion Criteria:

* Patients less than 15 years old as of the index date (<15 years old).
* Patients who were treated with 5-ASA during the baseline period (i.e. 12-month prior to the index date).
* Patients who were diagnosed with UC during the baseline period.
* Patients who received steroids, immunosuppressants, or biologics during the baseline period.

  * Steroid includes both oral medication and intravenous (IV) injection. The analysis will include the moderate- to high-dose of cumulative steroid use, which is defined as >=30mg of prednisolone, >= 50mg of methylprednisolone, or >=50mg of hydrocortisone.
  * Immunosuppressants is defined as at least one claim with Azathioprine or 6-Mercaptopurine.
  * Biologics is defined as at least one claim with Infliximab, Adalimumab, Ustekinumab, Vedolizumab, Golimumab, or Tofacitinib.
* Patients who were diagnosed with Crohn's disease at any time in the overall study period.

  * Defined as a claim with relevant Crohn's disease code recorded as primary diagnosis during the baseline period or follow-up period (i.e. entire study period).

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be selected from Korean HIRA claim database according to the inclusion/exclusion criteria. The Korean patients who were initially diagnosed with UC from 01 January 2009 to 30 June 2018 will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 11385 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Changes in initial 3-months average daily dose of 5-ASA | From prescription index date up to 3 months
  Initial average daily dose is defined as the average dose of 5-ASA prescribed over the 3-month period following the first prescription date of 5-ASA (i.e. prescription index date). Dose of 5-ASA includes those of mesalamine, sulfasalazine, and balsalazide.
  The dose will be stratified by oral monotherapy, rectal monotherapy, oral and rectal combination therapy. Oral and rectal combination therapy will be identified when the percentage of rectal therapy over the 3-months following the first prescription date of 5-ASA is more than 25%. For oral and rectal combination therapy, only oral formulation will be considered to calculate the dose of a combination therapy.
  The average daily dose of 5-ASA will be categorized as: Oral mono high dose (>=3g), oral mono standard dose (2-3g), oral mono low dose (<2g); Oral combination high dose (>=3g), oral combination standard dose (2-3g); oral combination low dose (<2g); Rectal monotherapy.
Prescription patterns of 5-ASA | From 01 January 2009 to 31 March 2019
  The prescription patterns will be categorized into: oral monotherapy; rectal monotherapy; oral and rectal combination therapy based on the exposure medications (mesalazine, sulfasalazine, and/or balsalazide) prescribed.

SECONDARY OUTCOMES:
Non-response to 5-ASA by the average daily dose of 5-ASA | From 01 January 2009 to 31 March 2019
  The non-response to 5-ASA is defined as: >=1 claims with international statistical classification of diseases 10th revision (ICD-10) code for UC as primary diagnosis and with pre-defined medications prescribed to those who are not responsive to 5-ASA. Medications for non-response are defined as add-on or switching to steroids, immunosuppressants, and/or biologics.
Ulcerative Colitis Related hospitalization by the average daily dose of 5-ASA | From 01 January 2009 to 31 March 2019
  The hospitalization is defined as: >=1 length of stay (days); admission to the department for gastroenterology; and at least one surgery code or UC medications. The UC surgery includes small bowel resection, colon resection, and/or low anterior resection, defined using surgery code. The UC medication is defined as moderate- to high-dose steroids, immunosuppressants, and/or biologics.
Ulcerative Colitis related surgery by the average daily dose of 5-ASA | From 01 January 2009 to 31 March 2019
  Surgeries include small bowel resection, colon resection, and/or low anterior resection, which will be identified using surgery code.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (1):
- Severance Hospital, Seoul, Seodaemun-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park SJ, Park SW, Cheon JH. Ten-Year Trend in 5-Aminosalicylic Acid Prescription Patterns and Treatment Outcomes in Patients with Ulcerative Colitis: An Analysis of Korean Health Insurance Data. Dig Dis Sci. 2025 Dec 23. doi: 10.1007/s10620-025-09629-0. Online ahead of print. PMID 41436897